CLINICAL TRIAL: NCT06253845
Title: A Phase 1b, Single Arm Study of CG0070 After Transurethral Resection in Patients With Intermediate Risk Non-Muscle Invasive Bladder Cancer (IR NMIBC)
Brief Title: Study of CG0070 After Transurethral Resection in Patients With IR NMIBC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21690
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Non-muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CG0070 (Experimental): CG0070 is a conditionally replicating oncolytic adenovirus (serotype 5) designed to preferentially replicate in and kill cancer cells.
  Interventions: Biological: CG0070

INTERVENTIONS:
Biological: CG0070 — CG0070 will be administered at a dose of 1x10^12 vp intravesically following a sequence of bladder washes with DDM and normal saline.

SUMMARY:
Investigators will evaluate the safety of CG0070 for the treatment of patients with Intermediate-Risk Non-Muscle Invasive Bladder Cancer (IR NMIBC).

ELIGIBILITY:
Inclusion Criteria:

* Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Have pathologically confirmed:

  * Recurrent Low-grade Ta
  * Solitary Low-Grade Ta > 3cm
  * Low-grade Ta multifocal
  * High-grade Ta ≤ 3cm
* Have all visible disease except a single "marker lesion" of approximately 0.3 - 1 cm diameter removed at baseline prior to initial CG0070 treatment (photographic documentation of lesion location and size must be conducted). "Marker lesion" must be clearly identifiable and assessable in the judgment of the investigator. "Marker lesion" location and size must be documented by the investigator (e.g., via photography).
* Demonstrate adequate organ function, defined as:

  * Aspartate transaminase (AST), alanine aminotransferase (ALT)

    ≤2.5 × upper limit of normal (ULN)
  * Total serum bilirubin ≤1.5 × ULN (OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN)
  * Absolute neutrophil count (ANC) ≥1,000 cells/mm3
  * Hemoglobin ≥8 g/dL or ≥4.96 mmol/L
  * Platelet count ≥100,000 platelets/mm3
  * Serum creatinine ≤1.5 × ULN or creatinine clearance ≥30 mL/min for patient with creatinine levels >1.5 institutional ULN according to Cockcroft-Gault formula
  * Serum chemistries: Sodium, potassium, and calcium within normal limits (WNL) or Grade 1
  * International normalized ratio (INR) or prothrombin time (PT) ≤1.5 × ULN unless receiving anticoagulation therapy and INR or PT is within the therapeutic range of intended use of anticoagulants. (NOTE: patients must be able to suspend, based on local practice, anticoagulant and anti-platelet therapy for study specific biopsies and procedures)
* Willing to use barrier contraception, as outlined in Section 6.6, during sexual activity, starting with Day 1 for up to 6 weeks after each dose of CG0070.
* Patients must be willing to comply with study mandated cystoscopies, urine cytology, CT urograms, biopsies, and other procedures (including transurethral resection of bladder tumor [TURBT] or other resection for all visible disease). Patients who withdraw consent for these procedures will be withdrawn from the trial.

Exclusion Criteria:

* Current or prior evidence of high-risk NMIBC defined as:

  * HG T1
  * Any recurrent HG (G3) Ta
  * HG Ta > 3 cm (or multifocal)
  * Any CIS
  * Any BCG exposure in HG patient
  * Any variant histology
  * Any LVI
  * Any HG prostatic urethral involvement
* Disease that is unable to be completely resected
* Lack of marker lesion
* Low-risk NMIBC defined as:

  * Low grade solitary Ta less than or equal to 3cm
  * Papillary urothelial neoplasm of low malignant potential
* Has current or past history of muscle invasive (T2 or higher stage) or locally advanced (T3/T4, any N) or metastatic bladder cancer
* Has history of high grade or low grade urothelial carcinoma in the upper genitourinary tract (kidneys, renal collecting systems, ureters) or prostatic urethra (including CIS of the urethra) within 12 months of enrollment
* Has received systemic anti-cancer therapy, including investigational agents, within 4 weeks of Day 1 NOTE: For participants who have entered the follow-up phase of an investigational study may participate if it has been 4 weeks after the last dose of the previous investigational agent
* Has any of the following within 6 months prior to starting study treatment: untreated myocardial infarction, untreated severe/unstable angina, coronary/peripheral artery bypass graft, cerebrovascular accident, pulmonary embolus, uncontrolled hypertension, or uncontrolled congestive heart failure that is deemed to be preventative from the patient completing study intervention and/or assessment.
* Has used excluded anti-viral medication (e.g., interferon/peg-interferon, ribavirin, etc.) within 14 days of Day 1 and that cannot be suspended throughout for at least 14 days prior to and after each treatment with CG0070. Please consult with sponsor to discuss any anti-viral that cannot be discontinued.
* Has had prior treatment with any human adenovirus serotype 5 based therapy (e.g., Ad-interferon or Adstiladrin/Instiladrin/nadofaragene firadenovec)
* Requires use of anti-platelet or anti-coagulant therapy that cannot be safely suspended for per protocol biopsies and other procedures as per standard of care
* Has significant immunodeficiency due to underlying illness (e.g., known HIV/AIDS). Note that HIV testing is not mandatory unless required by local health authorities.
* Has received systemic immunosuppressive medication including high-dose corticosteroids (e.g. systemic corticosteroids >10 mg prednisone or equivalent) within 28 days prior to Day 1. NOTE: Patients must not be receiving doses of >10 mg/day of prednisone or equivalent at the time of study entry or during the study and corticosteroids may not be used for premedication
* Has had an allogeneic tissue/solid organ transplant
* Has a known history of Hepatitis B (defined as HBsAg reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection
* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease
* Has a known additional malignancy that, in the opinion of the treating physician, may interfere with the study conduct or require on study treatment for the malignancy
* Has an active infection requiring systemic therapy (e.g., urinary tract infection or other active infection)
* Has received a live replication competent vaccine within 30 days prior to the first dose of study drug.
* Has not recovered (i.e., to ≤Grade 1 or to Baseline status) from AEs due to a previously administered agent or therapy
* Has an illness, metabolic dysfunction, physical examination finding, or clinical laboratory finding that gives reasonable suspicion of a disease or condition that would contraindicate study treatment or that would limit compliance with study requirements
* Is pregnant, currently breastfeeding or intending to breastfeed, within the projected duration of the trial beginning at Screening through 6 weeks after the last study treatment.
* IVE therapy within 8 weeks prior to beginning study treatment with the exception of cytotoxic agents (e.g., Mitomycin C, gemcitabine, doxorubicin, and epirubicin) when administered as a single instillation immediately following a TURBT procedure which is permitted up to 14 to 60 days prior to beginning study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Up to 2 years
  Adverse events Grade 3 or higher will be graded according to the NC Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.

SECONDARY OUTCOMES:
Complete Response Rate (CR) | 12 weeks
  CR as defined by the response assessment.
12-month recurrence free survival rate (RFS) | 12 months
  RFS is defined as the time from surgical removal of residual lesions after CG0070 treatment to recurrence of low- or high-grade urothelial carcinoma within the bladder.
24-month recurrence free survival rate (RFS) | 24 months
  RFS is defined as the time from surgical removal of residual lesions after CG0070 treatment to recurrence of low- or high-grade urothelial carcinoma within the bladder.
Progression free survival (PFS) | Up to 24 months
  PFS is defined as the time from documentation of Complete Response (CR) following CG0070 treatment to recurrence of low- or high-grade urothelial carcinoma within the bladder.
Cystectomy free survival (CFS) | Up to 24 months
  CFS is defined as the time from study registration to cystectomy performed for any cause. Reason for cystectomy will be collected and analyzed in conjunction with this endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Li, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States